CLINICAL TRIAL: NCT03265249
Title: Auricular Percutaneous Electrical Nerve Field Stimulation (PENFS) Using the BRIDGE Device for Post-Operative Pain Control in Patients Undergoing Liver Transplantation
Brief Title: BRIDGE Device for Post-operative Pain Control
Acronym: BRIDGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00084620
Record Dates: First submitted 2017-08-22; First posted 2017-08-29 (Actual); Results first posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-01

CONDITIONS: Liver Failure; Liver Diseases, Alcoholic; Liver Diseases; Pain, Postoperative; Transplant; Failure, Liver; Liver Cirrhosis, Biliary
MeSH Terms: conditions — Liver Failure; Liver Diseases, Alcoholic; Liver Diseases; Pain, Postoperative; Liver Cirrhosis, Biliary

STUDY DESIGN:
Intervention Model Description: Two groups where randomization is either to device or SOC (standard of care)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1 (Experimental): BRIDGE device will be placed prior to start of the surgery with standard of care pain control analgesia
  Interventions: Device: BRIDGE device
- Group 2 (No Intervention): Subjects will receive the standard of care pain control analgesia

INTERVENTIONS:
Device: BRIDGE device — an externally placed, FDA-cleared device that delivers percutaneous electrical stimulation with alternating frequencies to branches of cranial nerves (V, VII, IX, and X) through the external ear via a field effect
  Arms: Group 1

SUMMARY:
Auricular neurostimulation is a potential novel and non-invasive method of pain control following liver transplantation in a growing patient population with the probability of significant impact on economics and morbidity. The investigators propose a pilot study to investigate the effects of auricular neurostimulation in patients receiving a liver transplantation. The investigator will investigate the effects of auricular neurostimulation with this novel device and compare it to the current standard of care for pain management following liver transplantation.

DETAILED DESCRIPTION:
This is a prospective, randomized study to determine the efficacy of the BRIDGE device in reducing pain and opioid use in patients following liver transplantation. Subjects will be randomized in a 1:1 ration to one of the below groups:

Group 1: BRIDGE device will be placed prior to start of the surgery with standard of care pain control analgesia

Group 2: Subjects will receive the standard of care pain control analgesia

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  * ≥18 years of age but <70 years of age
  * Actively listed for isolated liver transplantation
  * Subject or legally authorized representative able to sign informed consent
  * Not currently treated with opioids or any medications that may interact with opioids
  * English speaking
  * Willing and able to participate and consent to this study

Exclusion Criteria:

* Diagnosis of acute liver failure or primary sclerosing cholangitis (PSC)
* Anticipated that the subject will require a new roux-en-y hepaticojejunostomy
* Current use of opioid use or other substance abuse.
* Chronic pain disorders
* Need for regional anesthesia (regional nerve blocks or epidurals)
* Adhesive allergy/sensitivity
* Subject admitted to the ICU at the time of transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Mavis, MD, Principal Investigator — Duke Universtity
Locations (1):
- Duke University, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- BRIDGE Device: BRIDGE device will be placed prior to start of the surgery with standard of care pain control analgesia
  BRIDGE device: an externally placed, FDA-cleared device that delivers percutaneous electrical stimulation with alternating frequencies to branches of cranial nerves (V, VII, IX, and X) through the external ear via a field effect
- Standard of Care: Subjects will receive the standard of care pain control analgesia
Period: Overall Study
Arm/Group | BRIDGE Device | Standard of Care
Started | 12 | 15
Completed | 12 | 14
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BRIDGE Device | Standard of Care | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.81 (10.17) | 55.98 (10.57) | 56.40 (10.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 7 | 11 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 15 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 9 | 15 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Opioid Usage After Surgery as Measured by Total Milligrams of Morphine or Equivalent (MEQ)
Time Frame: up to day 30
Measure: Mean (95% Confidence Interval); unit: milligrams morphine or equivalent (MEQ)
Arm/Group | BRIDGE Device | Standard of Care
Number analyzed (Participants) | 12 | 15
milligrams morphine or equivalent (MEQ) | 51.1 [36.6 to 65.6] | 45.4 [32.4 to 58.3]
Statistical Analysis 1: Comparison: BRIDGE Device vs Standard of Care; Test type: Superiority; p = 0.80, Mixed Models Analysis; Median Difference (Final Values) = 5.7, 95% CI 2-sided [-17.5 to 29]

2. Secondary Outcome: Pain Level
Description: Evaluation of the pain score in the two groups (SOC and with device) at the end of surgery
Time Frame: up to day 30
Reporting Status: Not Posted, anticipated posting 2023-09

3. Secondary Outcome: Reduction in Nausea Scores as Measured by a 4-item Questionnaire Response
Description: Determination of the intensity of nausea in the two groups (SOC and with device)
Time Frame: up to day 30
Reporting Status: Not Posted, anticipated posting 2023-09

4. Secondary Outcome: Reduction in Vomiting Scores as Measured by a 4-item Questionnaire Response
Description: Determination of the intensity of vomiting in the two groups (SOC and with device)
Time Frame: up to day 30
Reporting Status: Not Posted, anticipated posting 2023-09

5. Secondary Outcome: Reduction in Time for Return of Bowel Function as Measured by Length to Time of Bowel Functioning Return.
Description: Evaluation of return of bowel function noting day of bowel movement occurrence in both groups.
Time Frame: up to day 30
Reporting Status: Not Posted, anticipated posting 2023-09

6. Secondary Outcome: Incidence of Post-operative Ileus Will be Measured by Need for Nasogastric Decompression for >48 Hours
Description: Determination of the presence of an ileus in the two groups (SOC and with device)
Time Frame: up to 30 days
Reporting Status: Not Posted, anticipated posting 2023-09

7. Secondary Outcome: Improved Post-operative Mobility as Measured by the Patient Symptom Surveys
Description: Determination of mobility with in the two groups (SOC and with device)
Time Frame: up to 30 days
Reporting Status: Not Posted, anticipated posting 2023-09

8. Secondary Outcome: Reduction in Length of Hospital Stay as Measured by Days in Hospital
Description: Determination of length of hospital stay with in the two groups (SOC and with device)
Time Frame: up to 30 days
Reporting Status: Not Posted, anticipated posting 2023-09

ADVERSE EVENTS:
Time Frame: Up to 30 days
Arm/Group | BRIDGE Device | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 0/12 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/49/NCT03265249/Prot_SAP_000.pdf